CLINICAL TRIAL: NCT07045571
Title: Methylation Signature of Circulating Tumour DNA as a Prognostic and Theranostic Tool for Managing Pancreatic Ductal Adenocarcinoma
Brief Title: MSCAN: ctDNA Methylation as Prognostic and Theranostic Tool for Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: Yingbin Liu, MD, PhD, FACS (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Ruijin Hospital (Other); Changhai Hospital (Other)
Responsible Party: Sponsor-Investigator, Yingbin Liu, MD, PhD, FACS, principal investigator, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: PDAC_LB_2024
Record Dates: First submitted 2025-05-08; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Neoplasm; Pancreas Cancer
Keywords: Pancreatic ductal adenocarcinoma; Liquid biopsy; CtDNA; DNA methylation; Early diagnosis; Prognosis
MeSH Terms: conditions — Pancreatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- benign: benign pancreatic lesions
- malignant: malignant pancreatic lesions

SUMMARY:
Developing a characteristic ctDNA methylation panel for pancreatic ductal adenocarcinoma and establishing an intelligent diagnostic and dynamic monitoring model based on ctDNA methylation.

DETAILED DESCRIPTION:
Pancreatic cancer is a digestive system malignancy characterized by late clinical detection, high malignancy, and poor prognosis. Exploring economically viable, accurate, and minimally invasive methods for early diagnosis and postoperative monitoring is of significant clinical importance to facilitate early screening and improve patient outcomes. Liquid biopsy, which involves detecting various tumor-related biomarkers in extractable bodily fluids, such as circulating tumor cells, circulating tumor DNA, and exosomes, plays a crucial role in the early diagnosis and prognosis of pancreatic cancer.

Recent research indicates the substantial impact of liquid biopsy in the early diagnosis and prognosis of pancreatic cancer. Differential methylation regions in ctDNA, as opposed to ctDNA mutations, show promise as potential markers. Aberrant DNA methylation has been demonstrated to be more frequent than DNA mutations in tumor development and often occurs early in carcinogenesis. In this project, whole-genome methylation signal scans are conducted on blood samples and tumor tissue samples from pancreatic cancer using next-generation sequencing. The goal is to identify tumor-specific methylation biomarker sites. Subsequently, targeted sequencing is performed on ctDNA based on these identified sites.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting all inclusion criteria are eligible to enter this study, including but not limited to:

1. Age range between 18 and 80 years old;
2. Identification of pancreatic space-occupying lesions through imaging examinations, with a high suspicion of pancreatic malignant tumors and planned for surgical treatment or tissue biopsy for pathological confirmation;
3. According to RECIST 1.1 evaluation criteria, having at least one measurable lesion (the longest diameter of the target lesion on spiral CT scan ≥10mm);
4. Ability to provide tumor tissue and blood samples;
5. Stable vital signs, ECOG score of 0-1;
6. Liver function with AST and ALT ≤ 5 times the upper limit of normal (ULN), Child-Pugh classification of A or B; white blood cell count > 3×10^9/L, absolute neutrophil count ≥ 1.5×10^9/L; platelets ≥ 75×10^9/L; hemoglobin ≥ 90g/L; creatinine clearance rate ≥ 60ml/min; total bilirubin ≤ 3 times ULN;
7. Reproductive-age patients and their spouses willing to adopt contraceptive measures; female patients must undergo a pregnancy test (serum or urine) within 7 days before enrollment with a negative result.
8. Voluntarily participate in this experimental project, patients with good compliance; if the subject is unable to read or sign, the informed consent form must be signed by a legal representative with the subject's informed consent, and for subjects incapable of expressing consent, the introduction and explanation shall be provided to their legal representative, who will then sign the informed consent form.

Exclusion Criteria:

Patients meeting any of the exclusion criteria will not be eligible for inclusion, including but not limited to:

1. Unable to provide tumor tissue and blood samples;
2. Previously received molecular targeted therapy, immunotherapy, or anti-tumor radiochemotherapy before this study;
3. History of malignancies other than pancreatic malignancy;
4. Presence of other severe diseases, including but not limited to uncontrolled congestive heart failure (NYHA class III or IV), unstable angina, poorly controlled arrhythmias, uncontrolled moderate to severe hypertension (SBP > 160mmHg or DBP > 100mmHg);
5. Uncontrolled diabetes;
6. Active infection;
7. Patients with active autoimmune diseases requiring long-term use of steroids;
8. Patients who have undergone allogeneic transplantation;
9. Active psychiatric disorders affecting informed consent and/or protocol compliance;
10. Other severe illnesses deemed inappropriate for participation in this study by investigators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises individuals meeting inclusion criteria and not meeting any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of ctDNA in Early Screening for Pancreatic Cancer | Up to 2 years from start of study
  Measured using a targeted DNA methylation panel for ctDNA in plasma. The presence or absence of cancer will be confirmed by histopathological diagnosis. Sensitivity and specificity will be calculated using standard diagnostic test evaluation against the gold-standard diagnosis. "Early-stage" is defined as stage I or II pancreatic cancer confirmed by imaging and pathology.
Sensitivity and Specificity of ctDNA Methylation Test for Detection of Postoperative Recurrence | Up to 2 years from start of study
  Measured using plasma ctDNA methylation profiles collected at scheduled postoperative time points (e.g., every 3 months). Recurrence will be confirmed by imaging (CT/MRI) or biopsy when clinically indicated. Diagnostic accuracy (sensitivity/specificity) will be evaluated by comparing ctDNA results to confirmed recurrence status.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) Based on Imaging and Clinical Assessment | Up to 3 years from start of study
  PFS will be calculated from the date of enrollment to the date of disease progression or death from any cause. Disease progression will be assessed using RECIST 1.1 criteria via CT/MRI scans performed every 3-6 months.
Overall Survival (OS) | Up to 3 years from start of study
  Overall survival will be defined as the time from enrollment to death from any cause. Survival status will be monitored every 3 months through clinic visits or phone follow-up.
Early and Late Imaging Data | Up to 3 years from start of study
  CT and/or MRI imaging will be used to measure tumor size, vascular invasion, and metastasis at baseline and every 3-6 months. Data will be used to assess tumor response, progression, or recurrence.
Levels of Serum Tumor Biomarkers (CA19-9, CEA) in Early-Stage Pancreatic Cancer | Up to 3 years from start of study
  Serum levels of CA19-9 and CEA will be measured at baseline and during follow-up visits using standard immunoassays. Biomarker trends will be analyzed to assess correlation with disease stage, treatment response, and recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Yinbin Liu, PhD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Y, Seufert I, Al-Shaheri FN, Kurilov R, Bauer AS, Manoochehri M, Moskalev EA, Brors B, Tjaden C, Giese NA, Hackert T, Buchler MW, Hoheisel JD. DNA-methylation signature accurately differentiates pancreatic cancer from chronic pancreatitis in tissue and plasma. Gut. 2023 Nov 24;72(12):2344-2353. doi: 10.1136/gutjnl-2023-330155. PMID 37709492
- [Background] Garcia-Ortiz MV, Cano-Ramirez P, Toledano-Fonseca M, Aranda E, Rodriguez-Ariza A. Diagnosing and monitoring pancreatic cancer through cell-free DNA methylation: progress and prospects. Biomark Res. 2023 Oct 5;11(1):88. doi: 10.1186/s40364-023-00528-y. PMID 37798621